CLINICAL TRIAL: NCT01910636
Title: A Phase 3b, Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir Plus Ribavirin in Treatment-Naïve and Treatment-Experienced Japanese Subjects With Chronic Genotype 2 HCV Infection
Brief Title: Efficacy and Safety of Sofosbuvir Plus Ribavirin in Japanese Adults With Chronic Genotype 2 HCV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0118
Record Dates: First submitted 2013-07-23; First posted 2013-07-29 (Estimated); Results first posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis C
Keywords: HCV genotype 2 (GT-2)
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sofosbuvir+RBV 12 weeks (Experimental): Participants will receive sofosbuvir+RBV for 12 weeks.
  Interventions: Drug: Sofosbuvir; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg tablet administered orally once daily
  Other Names: GS-7977; PSI-7977; Sovaldi®
Drug: RBV — Ribavirin (RBV) tablets were administered orally in a divided daily dose according to package insert weight-based dosing according to the approved Copegus labeling in Japan (< 60 kg = 600 mg , > 60 kg to ≤ 80 kg = 800 mg, and ≥ 80 kg = 1000 mg)
  Other Names: Copegus®

SUMMARY:
This study will evaluate the antiviral efficacy, safety, and tolerability of sofosbuvir (SOF) plus ribavirin (RBV) in Japanese participants with chronic genotype 2 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Chronic genotype 2 HCV-infection
* Male or female, age ≥ 20 years
* Body weight ≥ 40 kg
* HCV RNA ≥ 10,000 IU/mL at screening

Exclusion Criteria:

* Current or prior history of clinically significant illness other than HCV
* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of a non-HCV etiology
* Infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Knox, Study Director — Gilead Sciences
Locations (19):
- Japan (19):
  - Akita
  - Chiba
  - Chiyoda-ku
  - Gifu
  - Ichikawa
  - Itabashi-ku
  - Izunokuni
  - Kita-ku
  - Kurashiki
  - Kurume
  - Matsumoto
  - Musashino
  - Nishinomiya
  - Ōgaki
  - Ōmura
  - Sapporo
  - Shinjuku-ku
  - Suita
  - Yamagata

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 20 study sites in Japan. The first participant was screened on 28 June 2013. The last study visit occurred on 09 June 2014.
Pre-assignment Details: 188 participants were screened.
Groups:
- SOF+RBV Treatment Naive: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (600-1000 mg daily based on weight) for 12 weeks (treatment naive)
- SOF+RBV Treatment Experienced: SOF 400 mg tablet once daily + RBV tablets (600-1000 mg daily based on weight) for 12 weeks (treatment experienced)
Period: Overall Study
Arm/Group | SOF+RBV Treatment Naive | SOF+RBV Treatment Experienced
Started | 90 | 63
Completed | 90 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug
Groups:
- SOF+RBV Treatment Naive: SOF 400 mg tablet once daily + RBV tablets (600-1000 mg daily based on weight) for 12 weeks (treatment naive)
- Total: Total of all reporting groups
Arm/Group | SOF+RBV Treatment Naive | SOF+RBV Treatment Experienced | Total
Number analyzed (Participants) | 90 | 63 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10.6) | 60 (8.8) | 57 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 26 | 83
  Male | 33 | 37 | 70
Cirrhosis Status [Number; unit: participants]
  No | 82 | 54 | 136
  Yes | 8 | 9 | 17
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 73 | 48 | 121
    CT | 17 | 11 | 28
    TT | 0 | 4 | 4
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.92) | 6.5 (0.66) | 6.3 (0.84)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 26 | 12 | 38
  ≥ 800,000 IU/mL | 64 | 51 | 115

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were enrolled, received at least 1 dose of study drug, and had chronic genotype 2 HCV infection.
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV Treatment Naive | SOF+RBV Treatment Experienced
Number analyzed (Participants) | 90 | 63
percentage of participants | 97.8 | 95.2

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation of Study Drug(s)
Description: The percentage of participants permanently discontinuing any study drug due to an adverse event was summarized.
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: participants who were enrolled and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- SOF+RBV: SOF 400 mg tablet once daily + RBV tablets (600-1000 mg daily based on weight) for 12 weeks
Arm/Group | SOF+RBV
Number analyzed (Participants) | 153
percentage of participants | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV Treatment Naive | SOF+RBV Treatment Experienced
Number analyzed (Participants) | 90 | 63
percentage of participants
  SVR4 | 98.9 | 95.2
  SVR24 | 97.8 | 95.2

4. Secondary Outcome: Percentage of Participants Experiencing Viral Breakthrough
Description: Viral breakthrough was defined as HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment, confirmed with 2 consecutive values (second confirmation value may have been posttreatment) or with a last available on-treatment measurement and no subsequent follow-up values.
Time Frame: Up to 12 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV Treatment Naive | SOF+RBV Treatment Experienced
Number analyzed (Participants) | 90 | 63
percentage of participants | 0 | 0

5. Secondary Outcome: Percentage of Participants Experiencing Viral Relapse
Description: Viral relapse was defined as having achieved undetectable HCV RNA levels (HCV RNA < LLOQ) at end of treatment, but did not achieve an SVR.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV Treatment Naive | SOF+RBV Treatment Experienced
Number analyzed (Participants) | 90 | 63
percentage of participants | 2.2 | 4.8

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF+RBV
Serious Adverse Events (participants affected / at risk) | 2/153
Other Adverse Events (participants affected / at risk) | 69/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (N=153)
Anaemia (Blood and lymphatic system disorders) | 1
Allergy to arthropod sting (Immune system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV (N=153)
Anaemia (Blood and lymphatic system disorders) | 18
Malaise (General disorders) | 11
Nasopharyngitis (Infections and infestations) | 45
Headache (Nervous system disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years